CLINICAL TRIAL: NCT02872558
Title: Shared Decision Making in Parents of Children With Acute Otitis Media: The Acute Otitis Media Choice Trial
Brief Title: Shared Decision Making in Parents of Children With Acute Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jana Anderson, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-000627
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Otitis Media Choice Decision Aid (Other): For patients whose clinician is randomized to the decision aid arm:
  1. The study coordinator will provide the decision aid for the parent/clinician dyad.
  2. The study coordinator will provide a color-printed copy of the decision aid to the clinician prior to the clinician having the antibiotics discussion with the parents.
  3. The study coordinator will offer to provide the treating clinician a concise refresher of the content included in the decision aid in the context of the trial.
  4. The clinician will then, using the decision aid as a tool to facilitate discussion regarding the natural course of AOM, pain control, antibiotics exposure and deeper infections.
  5. The clinician will then engage the parents in a shared decision regarding the use of immediate antibiotics versus a wait and watch prescription that is consistent with both the parent's values and preferences and the clinician's level of comfort.
  Interventions: Other: Acute Otitis Media Choice Decision Aid
- Usual Care (Other): the clinician will discuss management options with the parent in the clinician's usual fashion.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Acute Otitis Media Choice Decision Aid — Decision Aid
  Arms: Acute Otitis Media Choice Decision Aid
Other: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
This study will evaluate the efficacy of shared decision making in treatment of Acute Otitis Media in the Emergency Department setting.

DETAILED DESCRIPTION:
The Investigators long-term goal is to promote evidence-based, patient-centered evaluation in the acute care setting to more closely tailor antibiotic use to disease risk for Acute Otitis Media (AOM) in children.

The Investigator will conduct a single-center cluster randomized control trial comparing the efficacy, safety and patient-centered outcomes of the shared decision-making decision aid 'Acute Otitis Media Choice' to usual care among children diagnosed with acute otitis media in the ED for whom antibiotics are being considered to engage parents in shared decision-making.

ELIGIBILITY:
Inclusion:

1. 6 months to 18 years in age
2. Acute Otitis Media diagnosed (AOM) at the time of visit, defined as:

   * Middle Ear Effusion- demonstrated by pneumatic otoscopy, air fluid level, or a bulging tympanic membrane PLUS
   * Evidence of Acute Inflammation- opaque, white, yellow, or erythematous tympanic membrane or purulent effusion PLUS
   * Symptoms of otalgia, fussiness or fever

Exclusion:

1. Are currently on antibiotics
2. Have acute otitis media and another diagnoses that antibiotics are prescribed for
3. Have otitis-conjunctivitis syndrome
4. Have perforation of their tympanic membrane at time of diagnoses
5. Recurrent AOM defined as:

   1. ≥3 or greater separate AOM episodes in the previous 6 months or
   2. ≥4 or more greater AOM episodes in the previous 12 months with one in the last 6 months
6. Have a craniofacial abnormality
7. Have had previous ear tubes placed
8. Have an immunologic disorder
9. Are immunosuppression either by disease or medication
10. Are undergoing treatment for cancer :

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Number of parents completing the survey | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Anderson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson JL, Oliveira J E Silva L, Hess EP, Vanmeter DE, Mullan A, Brito JP, Hargraves IG, Bellolio F. Shared decision-making for pediatric acute otitis media in the United States: a randomized emergency department trial. BMC Emerg Med. 2025 Aug 2;25(1):146. doi: 10.1186/s12873-025-01305-w. PMID 40753428
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials